CLINICAL TRIAL: NCT03292926
Title: A Randomized Controlled Trial to Evaluate a Novel Analgesia Technique for ACL Reconstruction: Adductor Canal Block With an IPACK Versus Adductor Canal Block
Brief Title: A Novel Analgesia Technique for ACL Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-0934
Record Dates: First submitted 2017-09-20; First posted 2017-09-26 (Actual); Results first posted 2022-05-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Anterior Cruciate Ligament Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Bupivacaine; Ultrasonography; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adductor Canal Block (ACB) (Active Comparator): The adductor canal block will be ultrasound-guided sonosite. The anesthesiologist will administer 15 cc bupivacaine 0.5% with 2 mg preservative-free dexamethasone with a 22 gauge (G)/4 inch Chiba needle to the mid-thigh of the surgical limb while subject lays in the supine position post IV sedation.
  Interventions: Drug: Bupivacaine; Device: Ultrasound; Drug: Dexamethasone
- Adductor Canal Block & IPACK (ACB/IPACK) (Active Comparator): The adductor canal block will be ultrasound-guided. The anesthesiologist will administer 15 cc bupivacaine 0.5% with 2 mg preservative-free dexamethasone with a 22G/4 inch Chiba needle to the mid-thigh of the surgical limb while subject lays in the supine position post IV sedation.
  The IPACK will be ultrasound-guided with c60 sonosite probe (5-2Hz). While laying in the prone or supine, frog-leg position the IPACK will be administered using a 22G/4inch Chiba needle. The anesthesiologist will identify the popliteal artery at the popliteal crease and move cephalad just beyond the femoral condyles at the confluence with the femur. Then the anesthesiologist will identify the space between the femur and the popliteal artery and moving from medial to lateral place the needle in between the popliteal artery and femur with the tip ending 2-3 cm lateral to the artery and inject 25 cc bupivacaine 0.25% with 2 mg preservative-free dexamethasone.
  Interventions: Drug: Bupivacaine; Device: Ultrasound; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine will help treat pain and sensation after ACL repair
Device: Ultrasound — Ultrasound will guide anesthesiologist in performing the different nerve blocks
Drug: Dexamethasone — Dexamethasone will be used to prolong block duration
  Other Names: preservative free Dexamethasone

SUMMARY:
A comparison of two anesthetic techniques-- the Adductor Canal Block (ACB) and the Adductor Canal Block with Infiltration of the interspace between the popliteal artery and the capsule of the posterior knee (ACB/IPACK)-- in patients undergoing bone-tendon-bone (BTB) anterior cruciate ligament (ACL) reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing BTB ACL reconstruction with participating surgeon
* Age 13 or greater
* Planned use of regional anesthesia
* Ability to follow study protocol
* English speaking (secondary outcomes include questionnaires validated in English only)

Exclusion Criteria:

* Hepatic or renal insufficiency
* Younger than 13 years old
* Patients undergoing general anesthesia
* Allergy or intolerance to one of the study medications
* BMI > 40
* Diabetes
* American Society of Anesthesiology (ASA) score IV
* Chronic gabapentin/pregabalin use (regular use for longer than 3 months)
* Chronic opioid use (taking opioids for longer than 3 months, or daily morphine equivalent of >5mg/day for one month)
* Non-English speaking

Ages: 13 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Beathe, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Adductor Canal Block & IPACK (ACB/IPACK): The adductor canal block will be ultrasound-guided. The anesthesiologist will administer 15 cc bupivacaine 0.5% with 2 mg preservative-free dexamethasone with a 22G/4 inch Chiba needle to the mid-thigh of the surgical limb while subject lays in the supine position post IV sedation.
  The IPACK will be ultrasound-guided with c60 sonosite probe (5-2Hz). While laying in the prone or supine, frog-leg position the IPACK will be administered using a 22G/4inch Chiba needle. The anesthesiologist will identify the popliteal artery at the popliteal crease and move cephalad just beyond the femoral condyles at the confluence with the femur. Then the anesthesiologist will identify the space between the femur and the popliteal artery and moving from medial to lateral place the needle in between the popliteal artery and femur with the tip ending 2-3 cm lateral to the artery and inject 25 cc bupivacaine 0.25% with 2 mg preservative-free dexamethasone.
  Bupivacaine: Bupivacaine will help treat pain and sensation after ACL repair
  Ultrasound: Ultrasound will guide anesthesiologist in performing the different nerve blocks
  Dexamethasone: Dexamethasone will be used to prolong block duration
Period: Overall Study
Arm/Group | Adductor Canal Block (ACB) | Adductor Canal Block & IPACK (ACB/IPACK)
Started | 39 | 39
Completed | 39 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adductor Canal Block (ACB) | Adductor Canal Block & IPACK (ACB/IPACK) | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (7) | 25 (8) | 24 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 26 | 27 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 26 | 20 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 8 | 12
Region of Enrollment [Number; unit: participants]
  United States | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Pain While at Rest
Description: Average numerical rating scale (NRS) at rest. A lower score is a better outcome. scale ranges from 0 to 10.
Time Frame: 24 hours post-block administration
Population: some patients were lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adductor Canal Block (ACB) | Adductor Canal Block & IPACK (ACB/IPACK)
Number analyzed (Participants) | 37 | 37
score on a scale | 3.84 (1.86) | 3.95 (2.58)

2. Secondary Outcome: Discharge Criteria
Description: Time to meet discharge criteria utilizing the modified post anesthetic discharge scoring system. The frame represents when the measurements began, i.e. 3 hours after the administration of the anesthetic block. This represents time zero, at which recording would then begin.
Time Frame: From 3 hours post-block administration on Post-operative day (POD) 0 until met discharge criteria, assessed up to 1 day
Population: some patients lost to follow up
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Adductor Canal Block (ACB) | Adductor Canal Block & IPACK (ACB/IPACK)
Number analyzed (Participants) | 39 | 37
minutes | 180.67 (143.84) | 189.92 (254.55)

3. Secondary Outcome: Pain With Ambulation
Description: NRS Pain score with ambulation & stairs. A lower score is a better outcome. Score range is from 0 to 10.
Time Frame: 3 hours post-block administration on Post-operative day (POD) 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adductor Canal Block (ACB) | Adductor Canal Block & IPACK (ACB/IPACK)
Number analyzed (Participants) | 39 | 39
score on a scale
  NRS with Ambulation | 1.59 (1.43) | 1.26 (1.23)
  NRS with Stairs | 2.05 (1.92) | 2.1 (1.81)

ADVERSE EVENTS:
Time Frame: up to 7 days after surgery
Arm/Group | Adductor Canal Block (ACB) | Adductor Canal Block & IPACK (ACB/IPACK)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT03292926/Prot_SAP_000.pdf